CLINICAL TRIAL: NCT03297684
Title: Assessment of Biomarker Profile in Diabetic Macular Edema in Response to Treatment With Intravitreal Aflibercept
Brief Title: Assessment of Biomarker Profile in Diabetic Macular Edema With Intravitreal Aflibercept Injection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Advanced Eye Research Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: AERA101
Record Dates: First submitted 2017-09-27; First posted 2017-09-29 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aqueous humor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — Intravitreal injection aflibercept

SUMMARY:
To assess the biomarker profile in diabetic macular edema patients in response to intravitreal aflibercept injection. Patients with diabetic macular edema who meet study requirements will receive monthly intravitreal injections of aflibercept as approved by FDA for a period of 6 months. A small quantity of fluid will be removed from the vitreous at each injection for laboratory evaluation of biomarkers present before, during and after treatment with aflibercept.

DETAILED DESCRIPTION:
Study objective is to better understand the pathophysiology of diabetic macular edema (DME) by defining the factors that participate in the disease process or may be good biomarkers for disease progression. Study will investigate the temporal relationship between the course of treatment with anti-VEGF therapy and levels of candidate biomarkers previously identified to determine which biomarkers are affected by anti-VEGF therapy with aflibercept. Study will correlate response to therapy to particular biomarkers and attempt to identify those associated with resistance to therapy for DME. Biomarker data will be correlated with serial clinical evaluation of disease progression. 40 subjects with clinically significant DME who plan to undergo anti-VEGF therapy will be treated with intravitreal aflibercept monthly for 6 months. At each visit aqueous humor will be collected and stored (6 samples per patient). At termination of study all specimens will be analyzed for biomarkers identified from previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis type 1 or type 2 diabetes
* Clinical DME as assessed by OCT
* Well controlled glaucoma on medications but not on prostaglandin analogues
* Mild Age Related Macular Degeneration (AMD)
* Visual acuity between 73 and 5 ETDRS letters (20/40 -20/800 on eye chart)
* Willing and able to participate and to comply with clinic visits and procedures
* Provide signed informed consent

Exclusion Criteria:

* Unwillingness to participate or inability to understand or sign informed consent
* Poor eye fluid that would preclude adequate testing
* Prior intraocular treatment with anti-VEGF or focal laser treatment within 90 days
* Corticosteroid injections within 120 days
* Active proliferative diabetic retinopathy
* Intraocular pressure greater than 25 mm Hg
* Any previous vitrectomy surgery
* Current use of systemic anti-VEGF agents
* Shallow anterior eye chamber in eye with natural lens
* Non-diabetic related macular swelling (retinal vein occlusion)
* History of ocular disease
* Systemic disease other than diabetes mellitus
* Pregnant or breast feeding women
* Sexually active men or women of childbearing potential who are unwilling to practice adequate birth control during study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals with DME from the Dartmouth, MA geographic area who are patients of Advanced Eye Centers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure biomarkers in aqueous humor from individuals with DME | 2 years
  Identify temporal effects of treatment with intravitreal afflibercept

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Chatterton, MBA, JD, Study Director — Advanced Eye Research Associates
Locations (1):
- Advanced Eye Centers, South Dartmouth, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No